CLINICAL TRIAL: NCT01870791
Title: Phase II Trial of Palliative Epirubicin, Oxaliplatin & Capecitabine (EOX) Chemotherapy Combined With Omega-3 Fish Oil Infusion (Omegaven) in Patients With Oesophagogastric Carcinoma
Brief Title: Study of Additive Omega-3 Fish Oil to Palliative Chemotherapy to Treat Oesophagogastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11122; 2011-003950-24 (EudraCT Number)
Record Dates: First submitted 2013-05-28; First posted 2013-06-06 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Esophageal Neoplasm; Gastric Neoplasm
Keywords: Esophageal adenocarcinoma; Gastric adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — fish oil triglycerides; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omegaven (Experimental): Omegaven in combination with EOX chemotherapy
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Weekly omegaven infusion in combination with EOX chemotherapy
  Other Names: Omega-3 fish oil

SUMMARY:
The prognosis for patients with advanced oesophago-gastric cancer is poor. Approximately 16,000 patients in the United Kingdom die from the disease. In spite of new chemotherapy regimens, the average survival for these patients is around 9 months from diagnosis.

Omegaven is an infusion comprising omega-3 fish oils. There is evidence that omega-3 fish oil supplementation can improve general well-being and quality of life in patients receiving palliative chemotherapy for a number of different cancer types. It has also been suggested that omega-3 fish oil supplementation may reduce the toxicity of chemotherapy.

This clinical trial aims to see whether the addition of Omegaven to EOX chemotherapy, the most widely used regimen for patients with advanced oesophago-gastric cancer, will make this drug regimen more effective at killing oesophago-gastric cancer cells, such that disease progression is delayed. Forty-five patients who have been diagnosed with advanced oesophago-gastric cancer will be recruited over a two year period to receive standard chemotherapy and omega-3 fish oil supplementation. The results in these 45 patients will be compared to a matched historical control group of patients who have received identical chemotherapy. If results suggest that the combination of EOX and Omegaven is sufficiently effective, tolerable and feasible then it will be the intention of the trial team to take the combination forward to treat patients with advanced oesophago-gastric cancer in a randomised study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric or oesophageal carcinoma (irrespective of subtype), deemed incurable as a result of standard staging investigations.
* Measurable disease according to RECIST v1.1 criteria on CT within 4 weeks of study entry
* World Health Organization Performance status 0-2
* Aged >18 years
* Able to give informed written consent
* Life expectancy >12 weeks
* Adequate hepatic and renal function documented within 7 days prior to treatment (estimated glomerular filtration rate>50ml/min, serum bilirubin < 1.5x upper limit of normal; Alanine transaminase or aspartate transaminase < 2.5x upper limit of normal; Alkaline phosphatase< 3x upper limit of normal (in the absence of liver metastases). If liver metastases are present, serum transaminases < 5x upper limit of normal are permitted.)
* Adequate bone marrow function documented within 7 days (haemoglobin ≥9g/dL, platelets ≥100,000cells/mm3, neutrophil count ≥1500cells/mm3)
* Women of childbearing age must have a negative pregnancy test (urine or serum) at commencement of treatment
* Willing to use contraception if applicable
* Willingness to comply with scheduled visits, treatment, laboratory test, and other aspects of the trial

Exclusion Criteria:

* Prior radical treatment within 6 months of relapse
* Prior treatment with any systemic chemotherapy for metastatic disease
* Prior adjuvant radio- or chemotherapy within 4 weeks of starting the study
* Patients with locally advanced disease deemed suitable for radical chemo-radiotherapy
* Known hyperlipidaemic state
* Hypersensitivity to fish- or egg protein or to any of the active substances or constituents in the lipid emulsion
* Patients with known coagulation disorders
* Any general contra-indications to infusion therapy - pulmonary oedema, hyperhydration, decompensated cardiac insufficiency
* Any unstable medical conditions - uncontrolled diabetes mellitus, acute myocardial infarction, stroke, embolic disease, metabolic acidosis, sepsis, pancreatitis
* Known HIV or hepatitis B or C carrier
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with requirements of the protocol
* History of malignancy other than gastric or oesophageal cancer, with the exception of curative treatment for skin cancer (other than melanoma) or in situ breast or cervical carcinoma, or those treated with curative intent for any other cancer with no evidence of disease for 5 years
* Major surgical procedure or significant traumatic injury within 4 weeks of treatment
* Cerebral metastases
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan
* Known peripheral neuropathy > Grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible).
* Lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, or inability to take oral medication (administration of capecitabine by naso-gastric or jejunostomy feeding tube is permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Survival | 12 months
  Progression free survival from enrolment to disease progression

SECONDARY OUTCOMES:
Safety profile | 12 months
  The number of participants requiring dose delays
Efficacy | 6 and 12 months
  Objective response rate as assessed by RECIST v1.1
Safety profile | 12 months
  The number of participants experiencing adverse effects
Safety profile | 12 months
  The number of participants requiring dose modifications
Safety profile | 12 months
  The number of participants requiring treatment withdrawal due to adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: David J Bowrey, MD, Study Director — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Derived] Eltweri AM, Thomas AL, Fisk HL, Arshad A, Calder PC, Dennison AR, Bowrey DJ. Plasma and erythrocyte uptake of omega-3 fatty acids from an intravenous fish oil based lipid emulsion in patients with advanced oesophagogastric cancer. Clin Nutr. 2017 Jun;36(3):768-774. doi: 10.1016/j.clnu.2016.06.001. Epub 2016 Jun 7. PMID 27342748
- See also: European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-003950-24/GB